CLINICAL TRIAL: NCT02512380
Title: Neoadjuvant S1, Oxaliplatin, and Docetaxel (SLOT) Versus S1, Oxaliplatin(SOX) in Patients With Locally Advanced, Resectable Gastric/Esophagogastric Junction (EGJ) Cancer
Brief Title: Neoadjuvant SLOT Versus SOX in Patients With Locally Advanced, Resectable Gastric/Esophagogastric Junction (EGJ) Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Jing Huang, MD PhD, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CH-GI-069
Record Dates: First submitted 2015-07-29; First posted 2015-07-30 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-07

CONDITIONS: Gastric Adenocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SLOT group (Experimental): 4 cycles preoperative chemotherapy with Docetaxel+oxaliplatin+s1 . Gastric resection. 6 cycles adjuvant chemotherapy with sequential oxaliplatin+s1 or oxaliplatin+s1,then s1 for 6 months。
  Interventions: Drug: Docetaxel;oxaliplatin;s1
- SOX group (Active Comparator): 3 cycles preoperative chemotherapy with oxaliplatin+s1. Gastric resection. 4 cycles adjuvant chemotherapy with sequential oxaliplatin+s1
  Interventions: Drug: oxaliplatin;s1

INTERVENTIONS:
Drug: Docetaxel;oxaliplatin;s1 — Docetaxel 60mg/m2 was administered on day 1 of every 14 days.oxaliplatin 85 mg/m2 was administered on day 2 every 14 days. 40-60 mg of oral S-1 according to body-surface area twice a day was given for 10 days every 14 days .
  Arms: SLOT group
Drug: oxaliplatin;s1 — oxaliplatin 100 mg/m2 on day 1 every 21 days.40-60 mg of oral S-1 according to body-surface area twice a day was given for 2 weeks every 21 days .
  Arms: SOX group

SUMMARY:
gastric cancer is a highly aggressive malignancy with a poor overall outcome. The purpose of this study is to evaluate the 5-year survival of neoadjuvant S1, oxaliplatin, and docetaxel (SLOT) versus S1, oxaliplatin(SOX) in patients with locally advanced, resectable gastric/esophagogastric junction (EGJ) cancer.

DETAILED DESCRIPTION:
Two arms, phase 3 study of neoadjuvant S1, oxaliplatin, and docetaxel (SLOT) versus S1, oxaliplatin(SOX) in patients with locally advanced, resectable gastric/esophagogastric junction (EGJ) cancer. 380 Patients will be enrolled in this trial. The primary objective of this study is to determine the 5-year survival of the two arms.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven gastric or GE junction adenocarcinoma;
* Age: 18 to 70;
* ECOG 0-2;
* Adenocarcinoma of the stomach or GE junction according to staging classification TNM Scannographic: T3-4 N0/N + M0 ;
* Completion of baseline quality of life questionnaire
* Adequate bone marrow functions (ANC ≥ 1,500/ul, blood platelet ≥ 100,000/ul, haemoglobin ≥ 10g/dl);
* Adequate renal functions(serum creatinine ≤ 1.5mg/dl)
* liver functions (serum bilirubin ≤ 1.5UNL, AST/ALT ≤ 3 times(normal value)
* Written informed consent

Exclusion Criteria:

* Previous chemotherapy;
* Active infection requiring antibiotics
* Pregnant, lactating women
* Psychiatric illness, epileptic disorders
* Concurrent systemic illness not appropriate for chemotherapy
* History of other malignancy within 5 years except for non-melanoma skin cancer, cervix in situ carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Estimated)
Dates: Start 2015-07; Primary Completion 2019-07 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
5 year overall survival | 6 years

SECONDARY OUTCOMES:
3 year relapse free survival | 5 years
Surgical complete resection rate (R0) | 2.5 year
Pathological response rate | 2.5 year

OTHER OUTCOMES:
quality of life questionnaire | 6 year

CONTACTS AND LOCATIONS:
Overall Officials: Jing Huang, M.D., Study Chair — Cancer Hospital, CAMS
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, China